CLINICAL TRIAL: NCT00790218
Title: A Phase 1-2, Open-label, Dose-escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered CF102 in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Phase 1-2 Study of CF102 in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CF102-102HCC
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2022-05-17 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatoma; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — 2-chloro-N(6)-(3-iodobenzyl)adenosine-5'-N-methyluronamide

STUDY DESIGN:
Intervention Model Description: Study Arms: CF102 (1, 5, and 25 mg BID) in 28-day cycles.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CF102 1mg (Experimental): An open-label trial in 28-day cycles.
  Interventions: Drug: CF102
- CF102 5mg (Experimental): An open-label trial in 28-day cycles.
  Interventions: Drug: CF102
- CF102 25mg (Experimental): An open-label trial in 28-day cycles.
  Interventions: Drug: CF102

INTERVENTIONS:
Drug: CF102 — CF102 capsules twice daily by mouth
  Other Names: 2-Chloro-N6-(3-iodobenzyl)adenosine-5'-N-methyluronamide; Cl-IB-MECA

SUMMARY:
This trial will test the safety and efficacy of CF102 in patients with advanced liver cancer. Successive groups of patients will be given higher doses of CF102 by mouth on a twice-daily basis. Treatment will be assessed for adverse effects and for effects on the tumor.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-randomized, dose-escalation study, to be conducted in 2 phases: a dose-escalation phase, to determine the MTD of CF102 and to evaluate its safety/tolerability, PK, pharmacodynamic, and preliminary clinical activity; and a dose-confirmation phase, which will be a cohort expansion at or below the MTD (ie, the RP2D) of CF102. Subjects will be treated with oral doses of CF102 in consecutive, 28-day cycles. The initial dose of CF102 will be 1 mg twice daily (BID), with subsequent escalations to 5 and 25 mg BID, unless limited by toxicity. Subjects will be evaluated weekly for the first cycle, every 2 weeks for Cycles 2 and 3, and at the end of each subsequent cycle, up to 6 cycles of CF102 treatment. Subjects will return for a follow-up visit 28 days after completion of the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC:

   * For patients without underlying cirrhosis, diagnosis of HCC documented by cytology and/or histology
   * For patients with underlying cirrhosis, diagnosis of HCC established according to the American Association for the Study of Liver Diseases Practice Guideline algorithm (Appendix V).
2. HCC is advanced, refractory, or metastatic, and no standard therapies are expected to be curative.
3. At least 18 years of age.
4. For subjects in the dose-confirmation (RP2D) phase only: Measurable disease, using Response Evaluation Criteria in Solid Tumors (RECIST, Appendix IV). (Note that a lesion that has been subjected to radiotherapy or chemoembolization cannot be used as a target lesion.)
5. Eastern Collaborative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 at baseline.
6. The following laboratory values must be documented within 3 days prior to initiation of study drug:

   * Absolute neutrophil count (ANC) greater than or equal to 1 x 109/L
   * Platelet count greater than or equal to 50 x 109/L
   * Serum creatinine less than or equal to 2.0 mg/dL
   * Aspartic aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × upper limit of normal.
   * Total bilirubin ≤ 3.0 mg/dL.
   * Serum albumin ≥ 3.0 g/dL.
   * International normalized ratio (INR) ≤ 2.3.
7. Esophageal bleeding and varices, if present, have been sclerosed or banded, and no bleeding episodes have occurred during the prior 6 months.
8. Life expectancy of ≥ 12 weeks.
9. For women of childbearing potential, negative serum pregnancy test result.
10. Absence of active malignancy other than HCC within 2 years of entry, with the exception of basal cell carcinoma and squamous cell carcinoma of the skin.
11. Provide written informed consent to participate.
12. Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other study related procedures.

    -

Exclusion Criteria:

1. Any chemotherapy, immunomodulatory drug therapy, immunosuppressive therapy, corticosteroids > 20 mg/day prednisone or equivalent, or growth factor treatment (e.g., erythropoietin) within 14 days prior to initiation of study drug.
2. Major surgery or radiation therapy within 28 days prior to initiation of study drug.
3. Severe liver dysfunction (Child-Pugh Class C or hepatic encephalopathy).
4. Active infection requiring systemic therapy.
5. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
6. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females.
7. Pregnant or lactating female.
8. Women of childbearing potential, unless they agree to use dual contraceptive methods which, in the opinion of the Principal Investigator (PI), are effective and adequate for that patient's circumstances while on study drug.
9. Men who partner with a woman of childbearing potential, unless they agree to use effective, dual contraceptive methods (i.e., a condom, with female partner using oral, injectable, or barrier method) while on study drug.
10. Known human immunodeficiency virus- or acquired immunodeficiency syndrome-related illness.
11. Any severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the investigator's opinion, would make the patient inappropriate for entry into this study.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — Can-Fite BioPharma Ltd; Salomon Shtemmer, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Bar-Yehuda S, Stemmer SM, Madi L, Castel D, Ochaion A, Cohen S, Barer F, Zabutti A, Perez-Liz G, Del Valle L, Fishman P. The A3 adenosine receptor agonist CF102 induces apoptosis of hepatocellular carcinoma via de-regulation of the Wnt and NF-kappaB signal transduction pathways. Int J Oncol. 2008 Aug;33(2):287-95. PMID 18636149
- [Derived] Stemmer SM, Benjaminov O, Medalia G, Ciuraru NB, Silverman MH, Bar-Yehuda S, Fishman S, Harpaz Z, Farbstein M, Cohen S, Patoka R, Singer B, Kerns WD, Fishman P. CF102 for the treatment of hepatocellular carcinoma: a phase I/II, open-label, dose-escalation study. Oncologist. 2013;18(1):25-6. doi: 10.1634/theoncologist.2012-0211. Epub 2013 Jan 8. PMID 23299770
- See also: Can-Fite BioPharma Ltd — http://www.canfite.com

RESULTS

PARTICIPANT FLOW:
Groups:
- CF102 1mg; CF102 5mg; CF102 25mg: CF102: CF102 tablets were given orally twice daily
Period: Overall Study
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Started | 6 | 6 | 7
Completed | 5 | 6 | 7
Not Completed | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | CF102
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 12
Region of Enrollment [Number; unit: participants]
  Israel | 19

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Dose-limiting toxicity was defined as a clinically significant AE or laboratory abnormality occurring in Cycle 1
Time Frame: From start of treatment until Day 28 of Cycle 1
Population: Safety Population (all subjects receiving at least one dose of study drug)
Measure: Count of Participants; unit: Participants
Groups:
- CF102 1mg; CF102 5mg; CF102 25mg: CF102 tablets given orally, BID
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Number analyzed (Participants) | 6 | 6 | 7
Participants | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose
Description: The MTD was defined as the highest dose level at which < 2 of 6 patients developed Cycle 1 DLT.
Time Frame: first 28 days (Cycle 1)
Population: All subjects were evaluated for DLTs in the first cycle of therapy.
Measure: Number; unit: milligrams
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Number analyzed (Participants) | 6 | 6 | 5
milligrams | NA — No subjects in any cohort experienced dose-limiting toxicity, therefore analysis of maximum tolerated dose was not possible. | NA — No subjects in any cohort experienced dose-limiting toxicity, therefore analysis of maximum tolerated dose was not possible. | NA — No subjects in any cohort experienced dose-limiting toxicity, therefore analysis of maximum tolerated dose was not possible.

3. Primary Outcome: Maximum Plasma Concentration of CF102 (Cmax)
Description: Blood samples were collected and plasma concentrations determined using a high-pressure liquid chromatography method.
Time Frame: Dose Escalation Phase on Day 1 and Day 29 pre-dose and at 1, 2, 3, 4, 6, 8 hours post-dose
Population: The first 3 subjects in each dosing cohort participated in the pharmacokinetic sampling.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Number analyzed (Participants) | 3 | 3 | 3
ng/mL
  Day 1 | 4.455 (2.975) | 25.10 (16.93) | 98.36 (22.60)
  Day 29 | 10.46 (8.864) | 53.69 (31.76) | 330.6 (61.17)

4. Secondary Outcome: Number of Subjects With Objective Tumor Response
Description: Therapeutic effect of CF102 in hepatocellular carcinoma measured by number of subjects with objective tumor response
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Number analyzed (Participants) | 6 | 6 | 5
Participants | 0 | 0 | 0

5. Secondary Outcome: Relationship Between Biomarkers of Peripheral Blood Mononuclear Cell (PBMC) Adenosine A3 Receptor (A3AR) Expression and Clinical Effects of CF102
Description: The Peripheral Blood Mononuclear Cells (PBMC) were to be collected at Baseline and Day 28 in order to evaluate the Adenosine A3 receptor (A3AR) and PBMC biomarkers, and clinical effects of CF102.
Time Frame: Baseline to Day 28
Population: No data was collected for this exploratory endpoint.
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Over the course of the study to include. Up to 30 weeks (including up to 6 cycles of 28 days plus an approximately 30 day followup period).
Arm/Group | CF102 1mg | CF102 5mg | CF102 25mg
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/6 | 3/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF102 1mg (N=6) | CF102 5mg (N=6) | CF102 25mg (N=7)
Inflammation - knee (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hospitalization due to ascites paracentesis (Gastrointestinal disorders) | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 1
Fatigue (General disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
UTI (Infections and infestations) | 0 | 1 | 0
Thrombus - left leg (Vascular disorders) | 0 | 0 | 1
Pathological fracture sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF102 1mg (N=6) | CF102 5mg (N=6) | CF102 25mg (N=7)
Fatigue (General disorders) | 1 | 2 | 2
Asthenia (General disorders) | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pelvic pain (Gastrointestinal disorders) | 0 | 1 | 0
Petechiae (Blood and lymphatic system disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1
General Physical Health Deterioration (General disorders) | 1 | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Pathological Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No